CLINICAL TRIAL: NCT00634140
Title: Te Influence of Ezetimibe on Gallbladder Function
Brief Title: The Influence of Ezetimibe on Gallbladder Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated due to lack of funding support.
Sponsor: Indiana University (Other)
Responsible Party: Henry A. Pitt, MD, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0710-24
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Acalculous Cholecystitis
Keywords: gallbladder; ezetimibe for 4 to 6 weeks prior to gallbladder removal
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ezetimibe
  Interventions: Drug: ezetimibe
- 2 (Placebo Comparator): placebo for 4-6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10 mg daily for 4 to 6 weeks
  Other Names: Zetia
  Arms: 1
Drug: Placebo — placebo for 4-6 weeks
  Arms: 2

SUMMARY:
Ezetimibe is a drug which inhibits the absorption of both dietary and biliary cholesterol in the small intestine. Ezetimibe has been approved for use in humans to lower serum cholesterol.

The primary aim of this study is to determine if ezetimibe normalizes resting and residual volume in patients with chronic acalculous cholecystitis.

DETAILED DESCRIPTION:
Gallbladder disease continues to be a major healthcare problem in the United States with more than 750,000 cholecystectomies being performed each year. In the last decade, the proportion of elective cholecystectomies performed for chronic acalculous cholecystitis has more than doubled. During this same time, obesity has reached epidemic proportions. In addition, obesity-induced visceral steatosis is known to cause a local inflammatory process resulting in organ dysfunction, with nonalcoholic steatohepatitis being a well established example of this phenomenon. Previous data from our lab also have shown that both congenital and diet-induced obesity result in cholecystosteatosis, an increase in gallbladder wall fats accompanied by altered gallbladder motility and absorption. This phenomenon also has been documented in humans, with patients with chronic acalculous and/or calculous cholecystitis having increased gallbladder fat than nondiseased controls.

Ezetimibe is a drug which inhibits the absorption of both dietary and biliary cholesterol in the small intestine. Ezetimibe has been approved for use in humans to lower serum cholesterol. Moreover, ezetimibe has been shown to ameliorate hepatic steatosis and cholesterol gallstone formation in animal models. Previous data from our lab have documented that ezetimibe lowers serum cholesterol, prevents biliary crystals and ameliorates cholecystosteatosis in lean mice fed a high fat diet. However, the influence of ezetimibe on gallbladder motility, absorption and accumulation of toxic fats, metabolites, cytokines and chemokines, cholecystosteatosis, have not been studied in humans. Therefore, the aims of this study are 1) to determine if ezetimibe normalizes resting and residual volume in patients with chronic acalculous cholecystitis, 2) to determine if ezetimibe normalizes gallbladder ion flux in patients with chronic acalculous cholecystitis and 3) to determine if ezetimibe normalizes gallbladder absorption/secretion modulators as well as gallbladder fat, cytokines and chemkines.

Subjects with typical biliary pain and or ejection fraction less than 30% on a HIDA scan will be identified. Patients will then be randomized with one group given ezetimibe and the other group given placebo. All subjects will have gallbladder ultrasound studies to determine volume before and after a standardized fatty meal both before starting ezetimibe or placebo and after 4 weeks. A cholecystectomy will then be performed. In addition, pieces of the gallbladder taken at cholecystectomy will be analyzed for ion flux, as well as absorption/secretion modulators and accumulation of toxic fats, metabolites, cytokines and chemokines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with typical biliary pain and ejection fraction <30% on a HIDA scan.
* Must be > 18 years of age.

Exclusion Criteria:

* Subjects with gallstones seen on HIDA.
* Subjects on statin medication
* Subjects with known allergies to ezetimibe.
* Subjects who are pregnant or breast-feeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Normalization of resting gallbladder volume in patients with chronic acalculous cholecystitis | Approximately 6 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry A. Pitt, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States